CLINICAL TRIAL: NCT03076385
Title: A Phase 1, First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Immunogenicity of H10N8 Antigen mRNA in Healthy Adult Subjects
Brief Title: Safety, Tolerability, and Immunogenicity of VAL-506440 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAL-506440-P101; 2015-003452-48 (EudraCT Number)
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Influenza
Keywords: VAL-506440; H10N8 antigen mRNA; Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAL-506440 (Experimental)
  Interventions: Biological: VAL-506440
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAL-506440 — Escalating dose levels
  Arms: VAL-506440
Other: Placebo
  Arms: Placebo

SUMMARY:
This clinical study will assess the safety, tolerability and immunogenicity of VAL-506440 in healthy adult subjects.

ELIGIBILITY:
Inclusion

* Agrees to comply with the study procedures and provides written informed consent
* 18 to 64 years of age
* Body mass index between 18 and 30 kg/m2
* Negative urine pregnancy test at the Screening visit and the day of each vaccination.
* Female subjects must either be of non-childbearing potential or use highly effective methods of contraception from at least 2 months before the Screening Visit through 3 weeks post last vaccination
* In good health based on medical history, physical examination, vital sign measurements and laboratory safety tests performed prior to initial study vaccination

Exclusion

* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* Administration of an investigational product within 45 days
* Women who are pregnant or breastfeeding, or plan to become pregnant during the study
* Prior administration of investigational agent using formulations similar to VAL-506440
* History of a serious reaction to prior influenza vaccinations
* History of Guillain-Barré Syndrome within 6 weeks following a previous influenza vaccine
* Administration of any live attenuated vaccines within 4 weeks before enrollment, inactive vaccines within 2 weeks before enrollment, or plans to any vaccine within the vaccination period
* Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination
* Any chronic administration of immunosuppressant or other immune-modifying drugs within 6 months prior to administration of study vaccine
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
* Any acute disease at the time of enrollment
* Any bleeding risk or thromboembolic event or any related medical history
* Regular alcohol consumption > 3 units/day, or current user of any illicit drugs, or has a history of drug/alcohol abuse with 1 year of screening or has a positive urine drug/alcohol test at screening
* Persons employed in a capacity that involves handling poultry or wild birds
* Unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies within 4 weeks before administration of the first vaccination, throughout the study
* Had major surgery or donation of blood or blood products within 4 weeks of dosing
* Current smoking of more than 10 cigarettes (or equivalent amount of tobacco) per day, and within 3 months prior to Screening
* Subject is an employee of the Sponsor or CRO involved in the study.
* Vulnerable subjects (e.g., a subject kept in detention).
* Any condition, that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of the study results
* History of autoimmune disease
* Inadequate Liver Function as defined by AST, ALT, GGT, alkaline phosphatase and bilirubin > 1.5xULN
* Known allergy or history of anaphylaxis or other serious adverse reactions to any of the constituents of the study vaccine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 201 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Types, frequency, and severity of serious adverse events (SAE), adverse events of special interest (AESI), and adverse events considered related to study drug | Through 13 months of study participation

SECONDARY OUTCOMES:
Frequency of hemagglutinin inhibition (HAI) seroconversion measured by a neutralization assay in comparison with baseline samples | Through 13 months of study participation
Frequency of microneutralization seroconversion measured by a neutralization assay in comparison with baseline samples | Through 13 months of study participation

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feldman RA, Fuhr R, Smolenov I, Mick Ribeiro A, Panther L, Watson M, Senn JJ, Smith M, Almarsson Ӧ, Pujar HS, Laska ME, Thompson J, Zaks T, Ciaramella G. mRNA vaccines against H10N8 and H7N9 influenza viruses of pandemic potential are immunogenic and well tolerated in healthy adults in phase 1 randomized clinical trials. Vaccine. 2019 May 31;37(25):3326-3334. doi: 10.1016/j.vaccine.2019.04.074. Epub 2019 May 10. PMID 31079849